CLINICAL TRIAL: NCT02925403
Title: A Phase Ib Randomised, Controlled, Single-blind Study to Assess the Safety, Immunogenicity of the Malaria Vaccine Candidate R21 With Matrix-M1 Adjuvant in West African Adult Volunteers
Brief Title: A Study to Assess the Safety and Immunogenicity of the Malaria Vaccine, R21, With Matrix-M1 Adjuvant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC060
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2017-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group 1 (Active Comparator): 10μg R21/Matrix-M1 on days 0, 28, and 56.
  Interventions: Biological: R21/Matrix-M1
- Group 2 (Active Comparator): 50μg R21/Matrix-M1 on days 0, 28, and 56.
  Interventions: Biological: R21/Matrix-M1
- Group 3 (Placebo Comparator): Saline injection on days 0, 28, and 56.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: R21/Matrix-M1
  Arms: Group 1; Group 2
Other: Saline
  Arms: Group 3

SUMMARY:
This is a study in which healthy adult volunteers will be given either an experimental Malaria vaccine or a saline control vaccine.

Each volunteer will receive three vaccinations in total. Volunteers will be randomly allocated to one of two groups:

Group 1 will receive a low dose of the Malaria vaccine on days 0, 28, and 56. Group 2 will receive a saline solution on days 0, 28, and 56.

DETAILED DESCRIPTION:
A randomised, controlled, single-blind clinical trial to evaluate the safety and immunogenicity of the malaria vaccine candidate regime of three (3) doses of R21/Matrix-M1 compared with placebo, in healthy West African adult volunteers living in a malaria-endemic area.

The study will take place at the Centre National de Recherche et de Formation sur la Paludisme (CNRFP)/Unite de Recherche Clinique de Banfora (URC-B). Trial participants will be drawn from the Banfora Health Demographic system, which covers a total population of 30, 000.

Community sensitisation will be undertaken to engage the community with the study and recruit volunteers for participation in the study. The CNRFP study team will hold local community meetings and explain the study to the potentially eligible adult volunteers. During these meetings the investigators will explain the following: the need for a vaccine; the current status of vaccine development (including the fact that this is likely to be a prolonged process); the study screening and informed consent procedure; risks of vaccination and the unproven benefits of vaccination. It will be stressed that these are experimental vaccine regimens and cannot be guaranteed to provide protection, and that it will therefore still be necessary to seek treatment for possible malaria even after vaccination and they should continue to use other protective measures such as bed nets. It will be explained that to aid identification, a photograph of the volunteer will be taken if they are eligible to be enrolled in the trial.

After this meeting, based on the list of adults of suitable age for participation in the trial drawn from the DSS database, volunteers will be asked to participate in a public lottery that is made to randomly select participants who will be invited for a screening visit. All proposed volunteers thus selected will be invited to the Banfora clinical trials centre for the screening visit.

The Volunteer Information Sheet (VIS) will contain detailed information about the study and will be distributed to the proposed volunteers. The investigators will endeavour to ensure that all volunteers fully understand the risks. Any volunteer who appears to have less than complete understanding will be considered unable to give consent. If unable to sign, the volunteer will be asked to thumbprint the consent form in the presence of an impartial witness who will be present during the screening procedures and will countersign the consent form. Fully consented volunteers will undergo the full screening procedures. This consists of medical history, physical examination, and blood sampling for screening tests.

Volunteers will be randomised to receive either three (3) doses of R21/ Matrix-M1 or placebo (normal saline) as control. Simple randomisation into the study groups will be done by an independent statistician based at the University of Oxford. A randomisation code list will be generated by the independent statistician and its use guided by a clear Standard Operating Procedure (SOP). Allocation concealment will be employed by use of opaque sealed envelopes. As this is a single-blind clinical trial design, the laboratory scientists will be blinded to vaccine allocation until the end of the study.

Each volunteer will be monitored for one hour (or longer if necessary) after each vaccination. Each volunteer will be visited at home daily for 6 days after each vaccination (Days 0, 28, and 56) by a field worker for assessment and recording of any solicited and unsolicited AEs in diary cards. If necessary the volunteer will continue to be seen regularly until any observed AEs have resolved or stabilised. Scheduled visits at the CNRFP will be on Days 0, 7, 28, 35, 56, 63, 84, and 140. All volunteers will be followed up to Day 140 post-first vaccination for adverse events.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults ages 18 to 45 years.
* Willingness to remain in study area for the period of the study.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Women only: Must practice and show documented evidence of continuous effective contraception (e.g. depo-progesterone) or must be willing to take contraceptive measures not to become pregnant for the duration of the study. Willing to have pregnancy tests at screening and vaccination time points.
* Agreement to refrain from blood donation during the course of the study.
* Written informed consent to participate in the trial.

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Hb less than 10.0g/dl
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and chronic (more than 14 days) immunosuppressant or other immune-modifying drugs medication (for corticosteroids, this will mean prednisolone, or equivalent, ≥ 0.5mg/kg/day) within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or hypersensitivity reactions likely to be exacerbated by any component of the study vaccines.
* Any history of anaphylaxis post-vaccination.
* History of clinically significant contact dermititis.
* Pregnancy, lactation or intention to become pregnant during the study.
* Disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* History of splenectomy.
* Any other serious chronic illness requiring hospital specialist supervision.
* HIV or Hepatitis B surface antigen seropositivity.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat test will be requested.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred B Tiono, Principal Investigator — Centre National de Recherche et de Formation sur la Paludisme, Ouagadougou, Burkina Faso
Locations (1):
- Centre National de Recherche et de Formatation sur le Paludisme (CNRFP)/Unite de Recherche Clinique de Banfora (URC-B), Ouagadougou, Burkina Faso

REFERENCES:
- [Background] Sachs J, Malaney P. The economic and social burden of malaria. Nature. 2002 Feb 7;415(6872):680-5. doi: 10.1038/415680a. PMID 11832956
- [Background] Das P, Horton R. Malaria elimination: worthy, challenging, and just possible. Lancet. 2010 Nov 6;376(9752):1515-7. doi: 10.1016/S0140-6736(10)61551-6. Epub 2010 Oct 28. No abstract available. PMID 21035845
- [Background] White NJ. Antimalarial drug resistance. J Clin Invest. 2004 Apr;113(8):1084-92. doi: 10.1172/JCI21682. PMID 15085184
- [Background] Baird JK. Eliminating malaria--all of them. Lancet. 2010 Dec 4;376(9756):1883-5. doi: 10.1016/S0140-6736(10)61494-8. Epub 2010 Oct 28. No abstract available. PMID 21035840
- [Background] Alonso PL, Sacarlal J, Aponte JJ, Leach A, Macete E, Milman J, Mandomando I, Spiessens B, Guinovart C, Espasa M, Bassat Q, Aide P, Ofori-Anyinam O, Navia MM, Corachan S, Ceuppens M, Dubois MC, Demoitie MA, Dubovsky F, Menendez C, Tornieporth N, Ballou WR, Thompson R, Cohen J. Efficacy of the RTS,S/AS02A vaccine against Plasmodium falciparum infection and disease in young African children: randomised controlled trial. Lancet. 2004 Oct 16-22;364(9443):1411-20. doi: 10.1016/S0140-6736(04)17223-1. PMID 15488216
- [Background] Olotu A, Lusingu J, Leach A, Lievens M, Vekemans J, Msham S, Lang T, Gould J, Dubois MC, Jongert E, Vansadia P, Carter T, Njuguna P, Awuondo KO, Malabeja A, Abdul O, Gesase S, Mturi N, Drakeley CJ, Savarese B, Villafana T, Lapierre D, Ballou WR, Cohen J, Lemnge MM, Peshu N, Marsh K, Riley EM, von Seidlein L, Bejon P. Efficacy of RTS,S/AS01E malaria vaccine and exploratory analysis on anti-circumsporozoite antibody titres and protection in children aged 5-17 months in Kenya and Tanzania: a randomised controlled trial. Lancet Infect Dis. 2011 Feb;11(2):102-9. doi: 10.1016/S1473-3099(10)70262-0. Epub 2011 Jan 13. PMID 21237715
- [Background] RTS,S Clinical Trials Partnership; Agnandji ST, Lell B, Soulanoudjingar SS, Fernandes JF, Abossolo BP, Conzelmann C, Methogo BG, Doucka Y, Flamen A, Mordmuller B, Issifou S, Kremsner PG, Sacarlal J, Aide P, Lanaspa M, Aponte JJ, Nhamuave A, Quelhas D, Bassat Q, Mandjate S, Macete E, Alonso P, Abdulla S, Salim N, Juma O, Shomari M, Shubis K, Machera F, Hamad AS, Minja R, Mtoro A, Sykes A, Ahmed S, Urassa AM, Ali AM, Mwangoka G, Tanner M, Tinto H, D'Alessandro U, Sorgho H, Valea I, Tahita MC, Kabore W, Ouedraogo S, Sandrine Y, Guiguemde RT, Ouedraogo JB, Hamel MJ, Kariuki S, Odero C, Oneko M, Otieno K, Awino N, Omoto J, Williamson J, Muturi-Kioi V, Laserson KF, Slutsker L, Otieno W, Otieno L, Nekoye O, Gondi S, Otieno A, Ogutu B, Wasuna R, Owira V, Jones D, Onyango AA, Njuguna P, Chilengi R, Akoo P, Kerubo C, Gitaka J, Maingi C, Lang T, Olotu A, Tsofa B, Bejon P, Peshu N, Marsh K, Owusu-Agyei S, Asante KP, Osei-Kwakye K, Boahen O, Ayamba S, Kayan K, Owusu-Ofori R, Dosoo D, Asante I, Adjei G, Adjei G, Chandramohan D, Greenwood B, Lusingu J, Gesase S, Malabeja A, Abdul O, Kilavo H, Mahende C, Liheluka E, Lemnge M, Theander T, Drakeley C, Ansong D, Agbenyega T, Adjei S, Boateng HO, Rettig T, Bawa J, Sylverken J, Sambian D, Agyekum A, Owusu L, Martinson F, Hoffman I, Mvalo T, Kamthunzi P, Nkomo R, Msika A, Jumbe A, Chome N, Nyakuipa D, Chintedza J, Ballou WR, Bruls M, Cohen J, Guerra Y, Jongert E, Lapierre D, Leach A, Lievens M, Ofori-Anyinam O, Vekemans J, Carter T, Leboulleux D, Loucq C, Radford A, Savarese B, Schellenberg D, Sillman M, Vansadia P. First results of phase 3 trial of RTS,S/AS01 malaria vaccine in African children. N Engl J Med. 2011 Nov 17;365(20):1863-75. doi: 10.1056/NEJMoa1102287. Epub 2011 Oct 18. PMID 22007715
- [Background] Ewer KJ, O'Hara GA, Duncan CJ, Collins KA, Sheehy SH, Reyes-Sandoval A, Goodman AL, Edwards NJ, Elias SC, Halstead FD, Longley RJ, Rowland R, Poulton ID, Draper SJ, Blagborough AM, Berrie E, Moyle S, Williams N, Siani L, Folgori A, Colloca S, Sinden RE, Lawrie AM, Cortese R, Gilbert SC, Nicosia A, Hill AV. Protective CD8+ T-cell immunity to human malaria induced by chimpanzee adenovirus-MVA immunisation. Nat Commun. 2013;4:2836. doi: 10.1038/ncomms3836. PMID 24284865
- [Background] McConkey SJ, Reece WH, Moorthy VS, Webster D, Dunachie S, Butcher G, Vuola JM, Blanchard TJ, Gothard P, Watkins K, Hannan CM, Everaere S, Brown K, Kester KE, Cummings J, Williams J, Heppner DG, Pathan A, Flanagan K, Arulanantham N, Roberts MT, Roy M, Smith GL, Schneider J, Peto T, Sinden RE, Gilbert SC, Hill AV. Enhanced T-cell immunogenicity of plasmid DNA vaccines boosted by recombinant modified vaccinia virus Ankara in humans. Nat Med. 2003 Jun;9(6):729-35. doi: 10.1038/nm881. Epub 2003 May 25. PMID 12766765
- [Background] Webster DP, Dunachie S, Vuola JM, Berthoud T, Keating S, Laidlaw SM, McConkey SJ, Poulton I, Andrews L, Andersen RF, Bejon P, Butcher G, Sinden R, Skinner MA, Gilbert SC, Hill AV. Enhanced T cell-mediated protection against malaria in human challenges by using the recombinant poxviruses FP9 and modified vaccinia virus Ankara. Proc Natl Acad Sci U S A. 2005 Mar 29;102(13):4836-41. doi: 10.1073/pnas.0406381102. Epub 2005 Mar 21. PMID 15781866
- [Background] Nussenzweig RS, Vanderberg J, Most H, Orton C. Protective immunity produced by the injection of x-irradiated sporozoites of plasmodium berghei. Nature. 1967 Oct 14;216(5111):160-2. doi: 10.1038/216160a0. No abstract available. PMID 6057225
- [Background] Hill AV, Allsopp CE, Kwiatkowski D, Anstey NM, Twumasi P, Rowe PA, Bennett S, Brewster D, McMichael AJ, Greenwood BM. Common west African HLA antigens are associated with protection from severe malaria. Nature. 1991 Aug 15;352(6336):595-600. doi: 10.1038/352595a0. PMID 1865923
- [Background] Hill AV, Elvin J, Willis AC, Aidoo M, Allsopp CE, Gotch FM, Gao XM, Takiguchi M, Greenwood BM, Townsend AR, et al. Molecular analysis of the association of HLA-B53 and resistance to severe malaria. Nature. 1992 Dec 3;360(6403):434-9. doi: 10.1038/360434a0. PMID 1280333
- [Background] Todryk SM, Bejon P, Mwangi T, Plebanski M, Urban B, Marsh K, Hill AV, Flanagan KL. Correlation of memory T cell responses against TRAP with protection from clinical malaria, and CD4 CD25 high T cells with susceptibility in Kenyans. PLoS One. 2008 Apr 30;3(4):e2027. doi: 10.1371/journal.pone.0002027. PMID 18446217
- [Background] Khusmith S, Sedegah M, Hoffman SL. Complete protection against Plasmodium yoelii by adoptive transfer of a CD8+ cytotoxic T-cell clone recognizing sporozoite surface protein 2. Infect Immun. 1994 Jul;62(7):2979-83. doi: 10.1128/iai.62.7.2979-2983.1994. PMID 8005684
- [Background] Romero P, Maryanski JL, Corradin G, Nussenzweig RS, Nussenzweig V, Zavala F. Cloned cytotoxic T cells recognize an epitope in the circumsporozoite protein and protect against malaria. Nature. 1989 Sep 28;341(6240):323-6. doi: 10.1038/341323a0. PMID 2477703
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Background] Bejon P, Andrews L, Andersen RF, Dunachie S, Webster D, Walther M, Gilbert SC, Peto T, Hill AV. Calculation of liver-to-blood inocula, parasite growth rates, and preerythrocytic vaccine efficacy, from serial quantitative polymerase chain reaction studies of volunteers challenged with malaria sporozoites. J Infect Dis. 2005 Feb 15;191(4):619-26. doi: 10.1086/427243. Epub 2005 Jan 7. PMID 15655787
- [Background] Dunachie SJ, Walther M, Epstein JE, Keating S, Berthoud T, Andrews L, Andersen RF, Bejon P, Goonetilleke N, Poulton I, Webster DP, Butcher G, Watkins K, Sinden RE, Levine GL, Richie TL, Schneider J, Kaslow D, Gilbert SC, Carucci DJ, Hill AV. A DNA prime-modified vaccinia virus ankara boost vaccine encoding thrombospondin-related adhesion protein but not circumsporozoite protein partially protects healthy malaria-naive adults against Plasmodium falciparum sporozoite challenge. Infect Immun. 2006 Oct;74(10):5933-42. doi: 10.1128/IAI.00590-06. PMID 16988273
- [Background] Bejon P, Peshu N, Gilbert SC, Lowe BS, Molyneux CS, Forsdyke J, Lang T, Hill AV, Marsh K. Safety profile of the viral vectors of attenuated fowlpox strain FP9 and modified vaccinia virus Ankara recombinant for either of 2 preerythrocytic malaria antigens, ME-TRAP or the circumsporozoite protein, in children and adults in Kenya. Clin Infect Dis. 2006 Apr 15;42(8):1102-10. doi: 10.1086/501459. Epub 2006 Mar 14. PMID 16575727
- [Background] Bejon P, Mwacharo J, Kai OK, Todryk S, Keating S, Lang T, Gilbert SC, Peshu N, Marsh K, Hill AV. Immunogenicity of the candidate malaria vaccines FP9 and modified vaccinia virus Ankara encoding the pre-erythrocytic antigen ME-TRAP in 1-6 year old children in a malaria endemic area. Vaccine. 2006 May 29;24(22):4709-15. doi: 10.1016/j.vaccine.2006.03.029. Epub 2006 Mar 31. PMID 16621181
- [Background] Imoukhuede EB, Berthoud T, Milligan P, Bojang K, Ismaili J, Keating S, Nwakanma D, Keita S, Njie F, Sowe M, Todryk S, Laidlaw SM, Skinner MA, Lang T, Gilbert S, Greenwood BM, Hill AV. Safety and immunogenicity of the malaria candidate vaccines FP9 CS and MVA CS in adult Gambian men. Vaccine. 2006 Oct 30;24(42-43):6526-33. doi: 10.1016/j.vaccine.2006.06.022. Epub 2006 Jun 28. PMID 16842888
- [Background] Bejon P, Mwacharo J, Kai O, Mwangi T, Milligan P, Todryk S, Keating S, Lang T, Lowe B, Gikonyo C, Molyneux C, Fegan G, Gilbert SC, Peshu N, Marsh K, Hill AV. A phase 2b randomised trial of the candidate malaria vaccines FP9 ME-TRAP and MVA ME-TRAP among children in Kenya. PLoS Clin Trials. 2006 Oct 20;1(6):e29. doi: 10.1371/journal.pctr.0010029. PMID 17053830
- [Background] Keating SM, Bejon P, Berthoud T, Vuola JM, Todryk S, Webster DP, Dunachie SJ, Moorthy VS, McConkey SJ, Gilbert SC, Hill AV. Durable human memory T cells quantifiable by cultured enzyme-linked immunospot assays are induced by heterologous prime boost immunization and correlate with protection against malaria. J Immunol. 2005 Nov 1;175(9):5675-80. doi: 10.4049/jimmunol.175.9.5675. PMID 16237057
- [Background] O'Hara GA, Duncan CJ, Ewer KJ, Collins KA, Elias SC, Halstead FD, Goodman AL, Edwards NJ, Reyes-Sandoval A, Bird P, Rowland R, Sheehy SH, Poulton ID, Hutchings C, Todryk S, Andrews L, Folgori A, Berrie E, Moyle S, Nicosia A, Colloca S, Cortese R, Siani L, Lawrie AM, Gilbert SC, Hill AV. Clinical assessment of a recombinant simian adenovirus ChAd63: a potent new vaccine vector. J Infect Dis. 2012 Mar 1;205(5):772-81. doi: 10.1093/infdis/jir850. Epub 2012 Jan 24. PMID 22275401
- [Background] Ogwang C, Afolabi M, Kimani D, Jagne YJ, Sheehy SH, Bliss CM, Duncan CJ, Collins KA, Garcia Knight MA, Kimani E, Anagnostou NA, Berrie E, Moyle S, Gilbert SC, Spencer AJ, Soipei P, Mueller J, Okebe J, Colloca S, Cortese R, Viebig NK, Roberts R, Gantlett K, Lawrie AM, Nicosia A, Imoukhuede EB, Bejon P, Urban BC, Flanagan KL, Ewer KJ, Chilengi R, Hill AV, Bojang K. Safety and immunogenicity of heterologous prime-boost immunisation with Plasmodium falciparum malaria candidate vaccines, ChAd63 ME-TRAP and MVA ME-TRAP, in healthy Gambian and Kenyan adults. PLoS One. 2013;8(3):e57726. doi: 10.1371/journal.pone.0057726. Epub 2013 Mar 19. PMID 23526949
- [Background] Osman MM, Nour BY, Sedig MF, De Bes L, Babikir AM, Mohamedani AA, Mens PF. Informed decision-making before changing to RDT: a comparison of microscopy, rapid diagnostic test and molecular techniques for the diagnosis and identification of malaria parasites in Kassala, eastern Sudan. Trop Med Int Health. 2010 Dec;15(12):1442-8. doi: 10.1111/j.1365-3156.2010.02659.x. Epub 2010 Oct 25. PMID 20973878
- [Background] Rantala AM, Taylor SM, Trottman PA, Luntamo M, Mbewe B, Maleta K, Kulmala T, Ashorn P, Meshnick SR. Comparison of real-time PCR and microscopy for malaria parasite detection in Malawian pregnant women. Malar J. 2010 Oct 6;9:269. doi: 10.1186/1475-2875-9-269. PMID 20925928
- [Background] Imoukhuede EB, Andrews L, Milligan P, Berthoud T, Bojang K, Nwakanma D, Ismaili J, Buckee C, Njie F, Keita S, Sowe M, Lang T, Gilbert SC, Greenwood BM, Hill AV. Low-level malaria infections detected by a sensitive polymerase chain reaction assay and use of this technique in the evaluation of malaria vaccines in an endemic area. Am J Trop Med Hyg. 2007 Mar;76(3):486-93. PMID 17360872
- [Background] Bojang KA, Milligan PJ, Pinder M, Vigneron L, Alloueche A, Kester KE, Ballou WR, Conway DJ, Reece WH, Gothard P, Yamuah L, Delchambre M, Voss G, Greenwood BM, Hill A, McAdam KP, Tornieporth N, Cohen JD, Doherty T; RTS, S Malaria Vaccine Trial Team. Efficacy of RTS,S/AS02 malaria vaccine against Plasmodium falciparum infection in semi-immune adult men in The Gambia: a randomised trial. Lancet. 2001 Dec 8;358(9297):1927-34. doi: 10.1016/S0140-6736(01)06957-4. PMID 11747915
- [Background] Kester KE, Cummings JF, Ofori-Anyinam O, Ockenhouse CF, Krzych U, Moris P, Schwenk R, Nielsen RA, Debebe Z, Pinelis E, Juompan L, Williams J, Dowler M, Stewart VA, Wirtz RA, Dubois MC, Lievens M, Cohen J, Ballou WR, Heppner DG Jr; RTS,S Vaccine Evaluation Group. Randomized, double-blind, phase 2a trial of falciparum malaria vaccines RTS,S/AS01B and RTS,S/AS02A in malaria-naive adults: safety, efficacy, and immunologic associates of protection. J Infect Dis. 2009 Aug 1;200(3):337-46. doi: 10.1086/600120. PMID 19569965
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Background] Plebanski M, Gilbert SC, Schneider J, Hannan CM, Layton G, Blanchard T, Becker M, Smith G, Butcher G, Sinden RE, Hill AV. Protection from Plasmodium berghei infection by priming and boosting T cells to a single class I-restricted epitope with recombinant carriers suitable for human use. Eur J Immunol. 1998 Dec;28(12):4345-55. doi: 10.1002/(SICI)1521-4141(199812)28:123.0.CO;2-P. PMID 9862371
- [Background] Reece WH, Pinder M, Gothard PK, Milligan P, Bojang K, Doherty T, Plebanski M, Akinwunmi P, Everaere S, Watkins KR, Voss G, Tornieporth N, Alloueche A, Greenwood BM, Kester KE, McAdam KP, Cohen J, Hill AV. A CD4(+) T-cell immune response to a conserved epitope in the circumsporozoite protein correlates with protection from natural Plasmodium falciparum infection and disease. Nat Med. 2004 Apr;10(4):406-10. doi: 10.1038/nm1009. Epub 2004 Mar 14. PMID 15034567
- [Background] Schofield L, Villaquiran J, Ferreira A, Schellekens H, Nussenzweig R, Nussenzweig V. Gamma interferon, CD8+ T cells and antibodies required for immunity to malaria sporozoites. Nature. 1987 Dec 17-23;330(6149):664-6. doi: 10.1038/330664a0. PMID 3120015
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Tiono AB, Kangoye DT, Rehman AM, Kargougou DG, Kabore Y, Diarra A, Ouedraogo E, Nebie I, Ouedraogo A, Okech B, Milligan P, Sirima SB. Malaria incidence in children in South-West Burkina Faso: comparison of active and passive case detection methods. PLoS One. 2014 Jan 24;9(1):e86936. doi: 10.1371/journal.pone.0086936. eCollection 2014. PMID 24475198
- [Derived] Venkatraman N, Tiono AB, Bowyer G, Bellamy DG, Stockdale LK, Powlson J, Collins KA, Coulibaly S, Datoo MS, Silman D, Ouedraogo A, Nebie I, Imoukhuede EB, Brod F, Folegatti P, Dickinson-Craig E, Jamieson S, Bougouma EC, Wright D, Diarra A, Bliss CM, Morter R, Glenn G, Fries LF, Reimer JM, Lovgren-Bengtsson K, Baker M, Poulton I, Moyle S, Berrie E, Green N, Mukhopadhyay E, Viebig NK, Angus B, Lawrie A, Roberts R, Gilbert SC, Lewis DJM, Sirima SB, Ewer KJ, Hill AVS. Evaluation of a novel malaria anti-sporozoite vaccine candidate, R21 in Matrix-M adjuvant, in the UK and Burkina Faso: two phase 1, first-in-human trials. Lancet Microbe. 2025 Mar;6(3):100868. doi: 10.1016/S2666-5247(24)00084-3. Epub 2025 Jan 10. PMID 39805302

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 10μg R21/Matrix-M1 on days 0, 28, and 56.
  R21/Matrix-M1
- Group 2: Saline injection on days 0, 28, and 56.
  Saline
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 8 | 5
Completed | 8 | 4
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 5 | 0 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Administration of R21/Matrix-M1 Assessed by the Occurrence of Solicited Local and Systemic Adverse Events.
Description: Occurrence of solicited local and systemic adverse events (i.e: pain, redness, swelling and pruritus at injection site and temperature, feverishness, myalgia, arthralgia, malaise, headache and nausea).
Time Frame: Assessment of solicited AEs in the first 7 days post vaccination.
Measure: Number; unit: Number of adverse events
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 5
Number of adverse events | 10 | 0

2. Primary Outcome: Safety and Tolerability of R21/Matrix-M1 Assessed by the Occurrence of Unsolicited Adverse Events.
Description: Occurrence of unsolicited local and systemic adverse events. This will be done by recording the number of participants who experience unsolicited adverse events.
Time Frame: Unsolicited AEs to be assessed up to 28 days post vaccination.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 5
participants | 8 | 5

3. Primary Outcome: Safety and Tolerability of R21/Matrix-M1 Assessed by the Occurrence of Serious Adverse Events.
Description: Occurrence of serious adverse events will be collected from enrolment until the end of the follow-up period.
Time Frame: 6 months
Measure: Number; unit: SAEs
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 5
SAEs | 0 | 0

4. Primary Outcome: Safety and Tolerability of R21/Matrix-M1 Assessed by the Occurrence of Laboratory Adverse Events.
Description: Occurrence of laboratory adverse events defined as clinically significant changes from baseline. Haematology (Full Blood Count) and Biochemistry (Kidney and Liver Function Tests) will be assessed.
Time Frame: At Day 0 (baseline), day 7 and day 28 post vaccination.
Measure: Number; unit: Laboratory AEs
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 5
Laboratory AEs | 18 | 15

ADVERSE EVENTS:
Time Frame: Solicited adverse events will be recorded daily for 7 days post-vaccination Unsolicited AEs of all severities will be recorded from receipt of vaccination through 28 days post-vaccination. After study Day 28, only SAEs or new chronic medical conditions that require ongoing medical management will be recorded through to the last study visit.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=8) | Group 2 (N=5)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Vaccination 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Vaccination 1
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vaccination 1
Epigastralgia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vaccination 2
Ocular hyperhemia (Eye disorders) | 1 (1) | 0 (0) — Vaccination 3
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Vaccination 2
Furuncle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Vaccination 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Vaccination 3
Teeth decay (Infections and infestations) | 1 (1) | 0 (0) — Vaccination 1
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — Vaccination 1
Headache (General disorders) | 1 (1) | 0 (0) — Vaccination 1
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Vaccination 1
Neutropaenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) — Vaccination 1
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) — Vaccination 1
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Vaccination 2
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Vaccination 3
Neutropaenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) — Vaccination 2
Neutropaenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) — Vaccination 3
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) — Vaccination 2
Elevated Creatinine (Renal and urinary disorders) | 1 (1) | 1 (1) — Vaccination 3
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Vaccination 2
Swelling (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Vaccination 3
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Vaccination 3
Pain (General disorders) | 2 (2) | 0 (0) — Vaccination 1
Pain (General disorders) | 2 (2) | 0 (0) — Vaccination 2
Pain (General disorders) | 2 (2) | 0 (0) — Vaccination 3
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Vaccination 1
Headache (General disorders) | 2 (2) | 0 (0) — Vaccination 3
Headache (General disorders) | 2 (2) | 0 (0) — Vaccination 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Vaccination 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Vaccination 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Vaccination 3
Epigastralgia (Gastrointestinal disorders) | 1 (1) | 2 (2) — Vaccination 3
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) — Vaccination 2
Furuncle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Vaccination 2
Elevated ALT (Hepatobiliary disorders) | 0 (0) | 1 (1) — Vaccination 1
Elevated ALT (Hepatobiliary disorders) | 0 (0) | 1 (1) — Vaccination 2
Elevated ALT (Hepatobiliary disorders) | 0 (0) | 1 (1) — Vaccination 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT02925403/Prot_SAP_000.pdf